CLINICAL TRIAL: NCT01703741
Title: A Multicenter Extension Trial to Evaluate the Safety of FE 999303 (Testosterone Gel) in Adult Hypogonadal Males
Brief Title: A Multicenter Extension Trial to Evaluate the Safety of Testosterone Gel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000077
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Adult Male Hypogonadism
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone gel (FE 999093) (Experimental): Subjects received testosterone gel with initial dose as fixed on Day 56 (23 mg, 46 mg or 69 mg) during the 000023 study. The dose could further be down titrated based on serum testosterone levels at Day 90/91 of 000023 study. Testosterone gel was applied daily in morning using an applicator, to the shoulder/upper arm in a contralateral fashion for 6 months.
  Interventions: Drug: Testosterone Gel (FE 999093)

INTERVENTIONS:
Drug: Testosterone Gel (FE 999093)

SUMMARY:
This is a multicenter extension trial in adult hypogonadal males. The purpose of this study is to evaluate the safety of testosterone gel delivered using an applicator over an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the Phase 3 protocol (NCT01665599)

Exclusion Criteria:

* Use of another investigational product
* Use of any medications that could be considered anabolic or interfere with androgen metabolism
* Use of estrogens, gonadotropin releasing hormone agonists/antagonists, antiandrogens, or human growth hormone
* Use of another testosterone product
* Chronic use of any drug of abuse

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (18):
- United States (16):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - California Professional Research, Newport Beach, California
  - San Diego Sexual Medicine, San Diego, California
  - Connecticut Clinical Research, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Michigan Institute of Urology, Saint Clair Shores, Michigan
  - Premier Urology Associates, Lawrenceville, New Jersey
  - University Urology, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - PMG Research of Wilmington, Winston-Salem, North Carolina
  - Tristate Urologic Services, Cincinnati, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Clinical Research Associates, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
- Canada (2):
  - St. Joseph's Healthcare, London, Ontario
  - Private Practice and Clinical Research, North Bay, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 16 study centers in United States and 2 study centers in Canada.
Pre-assignment Details: Of the 172 subjects who completed study 000023 (NCT01665599), 145 subjects were enrolled into this extension study and continued to receive treatment (23 mg, 46 mg or 69 mg).
Groups:
- Testosterone Gel (FE 999303): Subjects received testosterone gel with initial dose as fixed on Day 56 (23 mg, 46 mg or 69 mg) during the 000023 study. The dose could further be down titrated based on serum testosterone levels at Day 90/91 of 000023 study. Testosterone gel was applied daily in morning using an applicator, to the shoulder/upper arm in a contralateral fashion for 6 months.
Period: Overall Study
Arm/Group | Testosterone Gel (FE 999303)
Started | 145
Per Protocol (PP) Population | 106 (Subjects having 24 hr pharmacokinetic (PK) data for testosterone, with no major protocol violations.)
Completed | 127
Not Completed | 18
Not completed — Withdrawal by Subject | 6
Not completed — Adverse Event | 2
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 3
Not completed — Subject did not want to continue | 2
Not completed — Subject cannot comply with study visits | 1
Not completed — Subject started testosterone injections | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population consists of all subjects who received at least one dose of Investigational Medicinal Product (IMP).
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 116
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 133
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 127
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Serum Total Testosterone Level - Maximum Observed Concentration (Cmax) of 1500-1799, 1800-2499, or Above 2500 ng/dL
Description: Measurement of total testosterone level occur after subjects have been on a stabilized dose of testosterone gel for at least one month in the period between Month 3 and Month 6.
  The data were presented using descriptive statistics.
Time Frame: Samples were collected at pre-dose; 2, 4, 6, 8, 10, 12 (±15 min for all), 18 (±2 hr), and 24 (±1 hr) hours post-dose (between Month 3 and Month 6, after subjects had been on a stabilized dose of Testosterone gel for at least 1 month)
Population: PP analysis population was used which comprises data from subjects who had 24 hr PK data for testosterone, with no major protocol violations.
Measure: Number; unit: percentage of subjects
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
percentage of subjects
  Total testosterone level between 1500-1799 ng/dL | 5.7
  Total testosterone level between 1800-2499 ng/dL | 2.8
  Total testosterone level above 2500 ng/dL | 2.8

2. Secondary Outcome: Percentage of Subjects With a Serum Total Testosterone Level (Average Steady State Concentration [Cave]) Between 300 and 1050 ng/dL.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
percentage of subjects | 82.1

3. Secondary Outcome: Domain Scores for the International Index of Erectile Function (IIEF) Questionnaire
Description: Data collected from the five domains of sexual functions were summarized by descriptive statistics.
  The domains are:
  1. Erectile function (6 items, questions 1-5 and 15) (Score range: 1-30)
  2. Orgasmic function (2 items, questions 9-10) (Score range: 0-10)
  3. Sexual desire (2 items, questions 11-12) (Score range: 2-10)
  4. Intercourse satisfaction (3 items, questions 6-8) (Score range: 0-15)
  5. Overall satisfaction (2 items, questions 13-14) (Score range: 2-10)
  A score of 0-5 is awarded to questions 1-10 and a score of 1-5 is awarded to questions 11-15. Low score indicates severe dysfunction and a high score indicates no dysfunction in sexual function, in each domain.
Time Frame: At Month 6
Population: ITT population was used which consists of all subjects who received at least one dose of the IMP. Of 145 treated subjects, 127 had available IIEF questionnaire results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 127
units on a scale
  Erectile function domain | 19.8 (7.9)
  Orgasmic function domain | 7.3 (3.2)
  Sexual desire domain | 7.0 (1.8)
  Intercourse satisfaction domain | 8.7 (4.4)
  Overall satisfaction domain | 6.7 (2.3)

4. Secondary Outcome: Percentage of Subjects With a Negative Androgen Deficiency in the Aging Male (ADAM) Questionnaire
Description: In ADAM questionnaire, subjects had to respond in "yes or no" to 10 questions. A positive result (with severity and symptoms of low testosterone) on the questionnaire was defined as an affirmative answer ("yes") to questions 1 or 7, or to any 3 other questions.
  The data were presented using descriptive statistics.
Time Frame: At Month 6
Population: ITT population was used which consists of all the subjects who received at least one dose of the IMP. Of 145 treated subjects, 127 had available ADAM questionnaire results.
Measure: Number; unit: percentage of subjects
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 127
percentage of subjects | 44.1

5. Secondary Outcome: Domain Scores for the Multidimensional Assessments of Fatigue (MAF) Questionnaire
Description: The MAF contains four sub-domains:
  1. Severity (2 items, questions 1-2) (Score range: 2-20)
  2. Distress (1 item, question 3) (Score range: 1-10)
  3. Degree of interference in activities of daily living (11 items, questions 4-14) (Score range: 11-110)
  4. Timing (2 items, questions 15-16) (Score range: 5-20)
  A score of 1-10 is awarded to each of the 14 questions across the 3 domains. The timing domain is categorical and was converted to 1-10 scale by multiplying each score by 2.5. Lower score in each domain indicates improvement in fatigue.
  To calculate GFI : Score of question 15 is converted to a 0-10 scale by multiplying each score by 2.5 and then sum scores of questions 1, 2, 3, average of 4-14, and newly scored question 15. A score of zero is assigned to question 2-16, if patient select 'no fatigue' to question 1. Question 16 is not included in GFI calculation. Range of GFI: 1 (no fatigue) to 50 (severe fatigue).
  The data were presented using descriptive statistics.
Time Frame: At Month 6
Population: ITT population was used which consists of all subjects who received at least one dose of the IMP. Of 145 treated subjects, 127 had available MAF questionnaire results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 127
units on a scale
  Severity domain | 6.6 (5.0)
  Distress domain: number analyzed (Participants) | 106
  Distress domain | 2.8 (2.3)
  Degree of interference in daily activities: number analyzed (Participants) | 107
  Degree of interference in daily activities | 28.3 (19.6)
  Timing domain: number analyzed (Participants) | 107
  Timing domain | 10.1 (3.2)
  Global fatigue index score | 15.3 (11.2)

6. Secondary Outcome: Domain Scores for the Short Form-12 (SF-12) Questionnaire
Description: Data collected from the SF-12 questionnaire was used to assess improvement in the psychometrically-based physical component summary (PCS) and mental component summary (MCS). Both PCS and MCS contains four sub-domains:
  PCS: General Health (1 item), Physical Functioning (2 items), Role-Physical (2 items), Bodily Pain (1 item)
  MCS: Role-Emotional (2 items), Mental Health (2 items), Vitality (1 item), Social Functioning (1 item)
  The scale scores are calculated by summing responses across scale items and then transforming these raw scores to a 0-100 scale. Computerized scoring algorithms are used to produce norm-based scores for each scale (mean of 50 and SD of 10) as well as the PCS and MCS summary scores. A zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
  The data were presented using descriptive statistics.
Time Frame: At Month 6
Population: ITT population was used which consists of all the subjects who received at least one dose of the IMP. Of 145 treated subjects, 127 had available SF-12 questionnaire results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 127
units on a scale
  General health domain | 54.3 (8.2)
  Physical functioning domain | 51.7 (8.6)
  Role-physical domain | 50.2 (8.4)
  Bodily pain domain | 51.1 (8.9)
  Physical component summary | 51.9 (8.1)
  Role-emotional domain | 48.8 (9.1)
  Mental health domain | 52.7 (8.0)
  Vitality domain | 53.1 (9.1)
  Social functioning domain | 51.2 (8.8)
  Mental component summary | 51.2 (8.3)

7. Secondary Outcome: Percentage of Subjects With a Serum Total Testosterone Level of 1500-1799, 1800-2499, or Above 2500 ng/dL
Description: The data were presented using descriptive statistics.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
percentage of subjects
  Total testosterone level between 1500-1799 ng/dL | 6.6
  Total testosterone level between 1800-2499 ng/dL | 5.7
  Total testosterone level above 2500 ng/dL | 2.8

8. Secondary Outcome: Percentage of Subjects With a Serum Total Testosterone Level of 1500-1799, 1800-2499, or Above 2500 ng/dL
Description: The data were presented using descriptive statistics.
Time Frame: At Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 105
percentage of subjects
  Total testosterone level between 1500-1799 ng/dL | 6.7
  Total testosterone level between 1800-2499 ng/dL | 2.9
  Total testosterone level above 2500 ng/dL | 1.9

9. Secondary Outcome: Area Under the Concentration-time Curve (AUCτ) for Total Testosterone and Dihydrotestosterone
Description: Measurement of total testosterone and DHT levels occur after subjects have been on a stabilized dose of Testosterone Gel for at least one month in the period between Month 3 and Month 6.
  The data were presented using descriptive statistics.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
ng*hr/dL
  Total testosterone at 23 mg: number analyzed (Participants) | 10
  Total testosterone at 23 mg | 7732 (1874)
  Total testosterone at 46 mg: number analyzed (Participants) | 40
  Total testosterone at 46 mg | 10583 (3863)
  Total testosterone at 69 mg: number analyzed (Participants) | 56
  Total testosterone at 69 mg | 10842 (3927)
  Total testosterone all doses | 10451 (3836)
  Dihydrotestosterone at 23 mg: number analyzed (Participants) | 10
  Dihydrotestosterone at 23 mg | 1361 (233)
  Dihydrotestosterone at 46 mg: number analyzed (Participants) | 40
  Dihydrotestosterone at 46 mg | 1675 (944)
  Dihydrotestosterone at 69 mg: number analyzed (Participants) | 56
  Dihydrotestosterone at 69 mg | 1751 (801)
  Dihydrotestosterone all doses | 1685 (827)

10. Secondary Outcome: Time at Which the Maximum Concentration (Tmax) Occurs for Total Testosterone and Dihydrotestosterone
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
hour
  Total testosterone at 23 mg: number analyzed (Participants) | 10
  Total testosterone at 23 mg | 3.09 [1.75 to 18.5]
  Total testosterone at 46 mg: number analyzed (Participants) | 40
  Total testosterone at 46 mg | 2.11 [0.0 to 24.1]
  Total testosterone at 69 mg: number analyzed (Participants) | 56
  Total testosterone at 69 mg | 3.97 [1.85 to 25.0]
  Total testosterone all doses | 3.88 [0.0 to 25.0]
  Dihydrotestosterone at 23 mg: number analyzed (Participants) | 10
  Dihydrotestosterone at 23 mg | 3.96 [0.0 to 24.9]
  Dihydrotestosterone at 46 mg: number analyzed (Participants) | 40
  Dihydrotestosterone at 46 mg | 4.00 [0.0 to 24.1]
  Dihydrotestosterone at 69 mg: number analyzed (Participants) | 56
  Dihydrotestosterone at 69 mg | 4.00 [0.0 to 25.0]
  Dihydrotestosterone all doses | 4.00 [0.0 to 25.0]

11. Secondary Outcome: Maximum Concentration Observed (Cmax) for Total Testosterone and Dihydrotestosterone
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
ng/dL
  Total testosterone at 23 mg: number analyzed (Participants) | 10
  Total testosterone at 23 mg | 747 (236)
  Total testosterone at 46 mg: number analyzed (Participants) | 40
  Total testosterone at 46 mg | 1085 (742)
  Total testosterone at 69 mg: number analyzed (Participants) | 56
  Total testosterone at 69 mg | 999 (525)
  Total testosterone all doses | 1008 (602)
  Dihydrotestosterone at 23 mg: number analyzed (Participants) | 10
  Dihydrotestosterone at 23 mg | 88.7 (21.0)
  Dihydrotestosterone at 46 mg: number analyzed (Participants) | 40
  Dihydrotestosterone at 46 mg | 111 (56)
  Dihydrotestosterone at 69 mg: number analyzed (Participants) | 56
  Dihydrotestosterone at 69 mg | 114 (62)
  Dihydrotestosterone all doses | 111 (57)

12. Secondary Outcome: Minimum Concentration Observed (Cmin) for Total Testosterone and Dihydrotestosterone
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
ng/dL
  Total testosterone at 23 mg: number analyzed (Participants) | 10
  Total testosterone at 23 mg | 162 (65)
  Total testosterone at 46 mg: number analyzed (Participants) | 40
  Total testosterone at 46 mg | 201 (98)
  Total testosterone at 69 mg: number analyzed (Participants) | 56
  Total testosterone at 69 mg | 219 (106)
  Total testosterone all doses | 207 (101)
  Dihydrotestosterone at 23 mg: number analyzed (Participants) | 10
  Dihydrotestosterone at 23 mg | 34.8 (7.5)
  Dihydrotestosterone at 46 mg: number analyzed (Participants) | 40
  Dihydrotestosterone at 46 mg | 43.5 (32.8)
  Dihydrotestosterone at 69 mg: number analyzed (Participants) | 56
  Dihydrotestosterone at 69 mg | 44.8 (26.9)
  Dihydrotestosterone all doses | 43.4 (28.1)

13. Secondary Outcome: Average Concentration (Cave) for Total Testosterone and Dihydrotestosterone
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Gel (FE 999303)
Number analyzed (Participants) | 106
ng/dL
  Total testosterone at 23 mg: number analyzed (Participants) | 10
  Total testosterone at 23 mg | 322 (78)
  Total testosterone at 46 mg: number analyzed (Participants) | 40
  Total testosterone at 46 mg | 438 (161)
  Total testosterone at 69 mg: number analyzed (Participants) | 56
  Total testosterone at 69 mg | 449 (165)
  Total testosterone all doses | 433 (160)
  Dihydrotestosterone at 23 mg: number analyzed (Participants) | 10
  Dihydrotestosterone at 23 mg | 56.6 (9.6)
  Dihydrotestosterone at 46 mg: number analyzed (Participants) | 40
  Dihydrotestosterone at 46 mg | 69.3 (39.5)
  Dihydrotestosterone at 69 mg: number analyzed (Participants) | 56
  Dihydrotestosterone at 69 mg | 72.4 (33.4)
  Dihydrotestosterone all doses | 69.7 (34.5)

ADVERSE EVENTS:
Time Frame: Overall study period (From Day 1 to Month 6)
Description: The treatment-emergent adverse event (TEAE), defined as any adverse event (AE) occurring after start of IMP administration and within the time of residual drug effect (5 days of the last dosing), or a pretreatment AE or pre-existing medical condition that worsens in intensity after treatment with the IMP and within the time of residual drug effect, were presented.
Groups:
- Testosterone Gel (FE 999303): Subjects received testosterone gel with initial dose as fixed on Day 56 during the 000023 study. The dose was further down titrated based on serum testosterone levels. Testosterone gel was applied using an applicator, to the shoulder/upper arm in a contralateral fashion.
Arm/Group | Testosterone Gel (FE 999303)
Serious Adverse Events (participants affected / at risk) | 1/145
Other Adverse Events (participants affected / at risk) | 28/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel (FE 999303) (N=145)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone Gel (FE 999303) (N=145)
Ventricular extrasystoles (Cardiac disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase abnormal (Investigations) | 1
Aspartate aminotransferase abnormal (Investigations) | 1
Haematocrit abnormal (Investigations) | 1
Haematocrit increased (Investigations) | 4
Haemoglobin abnormal (Investigations) | 1
Haemoglobin increased (Investigations) | 2
Red blood cell count abnormal (Investigations) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Presyncope (Nervous system disorders) | 1
Libido increased (Psychiatric disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 2
Epididymitis (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.